CLINICAL TRIAL: NCT02250820
Title: A Qualitative Comparison of Two Sedation Techniques in Children Undergoing Transthoracic Echocardiography
Brief Title: A Comparison of Two Sedation Techniques in Children Undergoing Transthoracic Echocardiography (TTE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2014-5961
Record Dates: First submitted 2014-09-16; First posted 2014-09-26 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Heart Disease
Keywords: Pediatric; Sedation; Transthoracic echocardiography; TTE; Dexmedetomidine; Pentobarbital
MeSH Terms: conditions — Heart Diseases | interventions — Dexmedetomidine; Pentobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal Dexmedetomidine and oral placebo (Experimental): If the patient is assigned to the dexmedetomidine arm, they will receive dexmedetomidine through the nose. In order to keep the assignment blinded, the patient will also receive an oral placebo.
  Interventions: Drug: Dexmedetomidine; Other: Oral Placebo
- Nasal placebo and oral pentobarbital (Experimental): If the patient is assigned to the pentobarbital arm, they will receive pentobarbital through the mouth. In order to keep the assignment blinded, the patient will also receive an nasal placebo.
  Interventions: Drug: Pentobarbital; Other: Nasal Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Nasal administration
  Arms: Nasal Dexmedetomidine and oral placebo
Drug: Pentobarbital — Oral administration
  Arms: Nasal placebo and oral pentobarbital
Other: Oral Placebo — Oral placebo will be cherry syrup
  Other Names: Cherry Syrup
  Arms: Nasal Dexmedetomidine and oral placebo
Other: Nasal Placebo — Nasal placebo will be nasally atomized saline
  Other Names: Nasally atomized saline
  Arms: Nasal placebo and oral pentobarbital

SUMMARY:
The study will examine the quality of two sedation techniques (dexmedetomidine and pentobarbital) used for children aged 3 to 24 months who are undergoing a transthoracic echocardiography (TTE).

DETAILED DESCRIPTION:
Currently there are two sedation methods used for children less than 24 months of age undergoing transthoracic echocardiography (TTE).

* One method provides sedation by mouth with the drug pentobarbital,
* The other provides sedation through the nose with the drug dexmedetomidine.

The choice of which method is used is based on evaluation of the patient's medical history and the preference of the anesthesiologist. To our knowledge, no study has compared these two sedation techniques for quality of care. The proposed study will help us determine which method yields the best quality and will allow us to improve the healthcare experience of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, scheduled to receive sedation for elective transthoracic echocardiography
* The subject must be a candidate for both anesthetic techniques. A staff member of the Division of Cardiac Anesthesiology will make this decision.
* The subjects must be 3 months to 24 months (inclusive of the 24th month).
* The subject's legally authorized representative has given written informed consent to participate in the study.

Exclusion Criteria:

* The subject has a history of cardiac conduction system disease (e.g. 1st or 2nd degree Atrioventricular block) or channelopathy (e.g. long QT syndrome).
* The subject is taking digoxin, alpha-adrenergic or beta-adrenergic agonist or antagonist (e.g., clonidine, propranolol, albuterol), anti-arrhythmic medications, or vasodilators (e.g. ACE inhibitors) on the day of the study procedures. It is routine for children taking these medications to hold them on the day of their procedure, as requested by the clinical team.
* The subject has received a dose of any other sedative within 48 hours.
* The subject has life-threatening, medical conditions (American Society of Anesthesiologists Physical Status 4, 5). The American Society of Anesthesiologists (ASA) classification scale is a measure of physical status or how healthy the patient is. For our study, we will focus on children which are defined as ASA I, II or III which means a healthy child (ASA I), a child with a systemic disease that is mild and well controlled (ASA II) or a child with systemic disease that is severe and controlled (ASA III).
* The subject is allergic to or has a contraindication to any of the drugs or masking flavored syrup used in the study.
* The subject has previously been treated under this protocol.
* The subject has Trisomy 21 (exaggerated risk of bradycardia)
* The subject has severe coarctation of the aorta (risk of exaggerated vasoconstriction)
* The subject has Moyamoya disease (risk of recurrent stroke)

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Sedation Quality | 60 minutes
  The primary outcome variable will be the sedation quality for the first 60 minutes after sedation drug is administered. It will be assessed if child is sedated within 30 minutes of administration of sedative drug, and if sedation is maintained for at least 30 minutes to allow a detailed transthoracic echocardiographic study. Sedation is defined as achieving Ramsay sedation level >3.

SECONDARY OUTCOMES:
Time to sedation | Participants will be followed for the time it takes to reach a sedated state, an expected average of 30 minutes
  Time from first dose of sedative medication to sedation. Sedation is defined as achieving Ramsay sedation level >3.
Delirium prior to sedation | Participants will be followed for the time it takes to reach a sedated state, an expected average of 30 minutes
  The incidence of delirium prior to achieving sedation.
Duration of sedation level >3 | Participants will be followed for the duration of the procedure, an expected average of 1 hour
Sonographer Pauses | Participants will be followed for the duration of the procedure, an expected average of 1 hour
  The number of sonographer pauses over 2 minutes due to patient movement or medical intervention will be counted.
Need for rescue nasal Dexmedetomidine | Participants will be followed for the duration of the procedure, an expected average of 1 hour
  The incidence of need for rescue nasal dexmedetomidine, due to patient arousal or movement prior to completion of TTE.
Incidence-severity of respiratory complications | Participants will be followed for the duration of their outpatient hospital stay, an expected average of 2 hours
  We will document the incidence and severity of respiratory complications (including supplemental oxygen).
Vital sign deviations of more than 30% from baseline | Participants will be followed for the duration of their outpatient hospital stay, an expected average of 2 hours
  We will document the incidence of blood pressure or heart rate deviations of more than 30% from baseline. Baseline will be measured prior to sedative administration.
Post anesthesia drowsiness or agitation | Participants will be followed for the duration of their post procedure stay, an expected average of 1 hour
  We will document the incidence-severity of post anesthesia drowsiness or agitation.
Duration of Post Anesthesia Care Unit (PACU) Phase | Participants will be followed for the duration of their post procedure stay, an expected average of 1 hour
  We will document the duration of stay in Post Anesthesia Care Unit (PACU) phase in minutes.
Time to oral fluid intake | Participants will be followed for the duration of their post procedure stay, an expected average of 1 hour
  We will document the time (in minutes) to oral fluid intake during the PACU phase
Time to discharge | Participants will be followed for the duration of their post procedure stay, an expected average of 1 hour
  We will document the time it takes a patient to be discharged from the hospital after the completion of the TTE.
Satisfaction of the Parents | up to 3 days
  The satisfaction of the sedation technique will be completed by the parents by asking a series of questions during a follow-up phone call the next business day after the TTE.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Miller, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Miller JW, Ding L, Gunter JB, Lam JE, Lin EP, Paquin JR, Li BL, Spaeth JP, Kreeger RN, Divanovic A, Mahmoud M, Loepke AW. Comparison of Intranasal Dexmedetomidine and Oral Pentobarbital Sedation for Transthoracic Echocardiography in Infants and Toddlers: A Prospective, Randomized, Double-Blind Trial. Anesth Analg. 2018 Jun;126(6):2009-2016. doi: 10.1213/ANE.0000000000002791. PMID 29369091